CLINICAL TRIAL: NCT03605615
Title: VocalizationTechnique During the Second Period of Labor Versus Usual Care for Prevention of Perineal Trauma: Randomized Clinical Trial
Brief Title: Vocalization for the Second Stage of Labor (VOCAL)
Acronym: VOCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, Principal Investigator, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VOCAL
Record Dates: First submitted 2018-07-09; First posted 2018-07-30 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Perineal Tear; Perineum; Rupture
Keywords: vaginal delivery; perineal tear; randomized controled trial
MeSH Terms: conditions — Rupture | interventions — Singing

STUDY DESIGN:
Intervention Model Description: This will be a randomized open-label trial with the objective of evaluating the effect of vocalization as a perineal protection maneuver during the second stage of labor. Paerturients will be randomized to receive standard care, which in the ward is already a humanized approach, with freedom of position, and to push, ou to, toguether with all this standard prodedure, receive orientation about vocalization techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): In this group parturients will be attended in standardized manner, which in our hospital means a humanized approach with choice of position in socond stage and without routine episiotomy.
- VOCALIZATION (Experimental): In this group parturients will besides being be attended with our standar care, will receive training to vocalize during second stage.
  Interventions: Other: vocalization

INTERVENTIONS:
Other: vocalization — The vocalization will be taught in voice form exhaled / sung in grave tones with the vowels, A, O and U.
  Other Names: vocalization technique; open glottis
  Arms: VOCALIZATION

SUMMARY:
A randomized open-label trial will be conducted to evaluate the effect of vocalization as a perineal protection maneuver during the second period of labor. The study will be carried out in the "Espaço Aconchego" sector of the IMIP, which has a team of obstetrical nurses, medical coordination and physiotherapeutic support. The study population will consist of low-risk parturients, with no prior cesarean indication, admitted to the sector. Those parturients who meet the inclusion criteria, after signing the Informed Consent Term, will be allocated to two groups: Group A (experimental) and Group B (control). Group A will be stimulated to keep the glottis minimally open during spontaneous pushing and to emit sounds when exhaling (vocalization), and Group B will undergo usual routine. Study outcomes will be evaluated by assistents immediately after delivery. After 24 hours of delivery, the conditions of the perineum will be assessed by inspection and palpation of the region,evaluating the presence of edema or other abnormality.

DETAILED DESCRIPTION:
SAMPLE SIZE As there are no studies to perform an adequate sample calculation, the present study will consist of 40 women, randomly randomized to use or not the vocalization technique, 20 in each group ( pilot exploratory study).

SAMPLING Sampling shall be obtained for convenience, consecutively.

Low-risk pregnant women admitted to the "Espaço Aconchego" sector who meet the eligibility criteria, will be questioned by the researcher about the interest in participating in the study in question. The objective of the vocalization technique will be explained to the pregnant woman, with the main aim being the prevention of perineal laceration and the probable prevention of postpartum complaints. In the case of parturients above 18 years, the Free and Informed Consent Form will be given and will be read and explained aloud, and only those who freely agree to participate, signing the term, will be included in the survey. In the case of under-age parturients, the legal guardians will sign the Informed Consent.

VARIABLE DEFINITIONS

Perineal laceration: categorical variable, involving two categories:

* Present - when there is some degree of solution of continuity of the skin or mucosa in the posterior region of the perineum, which reaches or not the subcutaneous and the muscle.
* Absent - defined as the posterior region of the intact perineum, without any solution of tissue continuity.

Duration of the active delivery period: numerical variable, determined in minutes (min), from total dilatation of the uterine cervix to the complete exit of the fetus associated with the spontaneous pull performed by the woman.

The degree of laceration will be classified according to the damaged tissues and defined according to the following criteria:

* First degree laceration: involves the skin, the subcutaneous tissue and the vaginal mucosa or the combination of multiple superficial lacerations, reaching the tissues already mentioned;
* Second degree laceration: involves the superficial muscles (bulbocavernosus and transverse); if it is deep, it also reaches the pubococcygeus muscle;
* Third degree laceration: involves the set of superficial and deep muscles of the anal sphincter:
* Fourth degree laceration: involves the set of muscles of the anal sphincter and the anal epithelium.

Location of vulvoperineal laceration

* Anterior region: clitoris, small left lip, small right lip, left vestibular region and right vestibular region;
* Posterior region: corresponding to the perineum itself (left side, right side and median region).

Size of laceration: extension in centimeters of perineal laceration; continuous numeric variable; Need for perineal suture: dichotomous categorical variable type (yes / no), expressed according to the need for perineal suture; Number of threads used for perineal suture: discrete numerical variable, corresponding to the number of threads partially or totally used for the suture of perineal lacerations; Use of oxytocin after randomization: dichotomous categorical variable (yes / no), defined by the placement or not of the hormone at the time of delivery, after randomization; Episiotomy: dichotomous categorical variable type (yes / no), defined as a surgical incision performed on the perineum at the time of vaginal delivery; Instrumental delivery: dichotomous categorical variable type (yes / no), after leasing of the forceps or vacuum-extractor, followed by elevation of the cephalic pole, if considered necessary; Perineal edema: dichotomous categorical variable type (yes / no), defined as fluid accumulation in the interstitium of perineal tissues by subjective evaluation of the examiner.66 Perineal Pain through the Visual Analogue Scale (EVA): continuous variable, describing the level of pain referred by the patient at each evaluation, ranging from zero to ten, with zero being the total absence of pain and ten the most extreme pain, unbearable, never felt in the course of life67 Maternal satisfaction: Categorical ordinal variable determining the level of maternal satisfaction after delivery. They will be considered satisfied, very satisfied, dissatisfied and not very satisfied.

Apgar scores of the newborn: continuous numerical variable, corresponding to the Apgar score recorded in the first and fifth minutes after birth, performed by the neonatologist, categorized as: 1 min ≥ 7, 1 min <7, 5 min ≥ 7, 5th min <7.

Need of resuscitation: categorical variable yes / no corresponding to the need for resuscitation of the baby after delivery from the PPV or larger interventions.

Neonatal ICU need: categorical variable type yes / no corresponding to the need for neonatal ICU, categorized as: yes or no.

Spontaneous Pushing: when performed without interference of the team assisting the parturient; Guided Guidance: when performed with interference from the team that assists the woman patient; Maternal Age: variable expressed in complete years, according to the patient's information, at the moment of data collection; Weight: Continuous numerical variable (which can later be categorized), expressed in kilos, indicating the weight of the patient at the moment of the study. Information collected by the patient's medical record; Height: Continuous numerical variable (can be later categorized), expressed in meters, indicating its height. Information collected from the medical records at the time of their selection to enter the study; BMI: continuous numerical variable, which represents the woman's body mass index. The formula for arriving at this value is weight / height²; Schooling: categorical variable informed by the patient and categorized as illiterate, high school, elementary school, higher education; Conjugal situation: categorical and police variables reported by the patient with or without a partner; Occupation: categorical variable informed by the patient; Kristeller's maneuver: dichotomous categorical variable, type yes / no, defining whether the parturient received some fundal pressure performed by the obstetric team. You will be informed by someone from the team who attended the delivery that saw the birth; Valsalva maneuver> six seconds: dichotomous categorical variable, yes / no type, indicating if the woman was instructed to perform forces contracting her perineal muscles and holding her breath at the moment of uterine contractions; Number of pregnancies: discrete variable. Expressed by the number of times the pregnant woman became pregnant, including the current gestation; Number of births: a discrete numerical variable, corresponding to the number of births (birth after 20 weeks or newborn weight greater than or equal to 500 grams), according to the patient's or family members' information; Gestational Age in Weeks: continuous variable, recorded as discrete, recorded in full weeks obtained preferably from the date of the last menstruation (LMP) or by ultrasonography; Newborn weight: numerical variable measured by the weight of the newborn in grams (g) immediately after birth; Cephalic perimeter of the Newborn: numerical variable measured in centimeters (cm) of the newborn's head circumference.

The statistical analysis will be carried out by the researchers, in addition to the statistician involved in the research, using the statistical programs Epi-Info 3.5.4 The statistical analysis will be performed with the groups identified as A or B, breaking the confidentiality only after obtaining the results and prepared tables. Thus, it will only be known which group was oriented on vocalization or not at the end of the analysis.

Categorical variables will be compared in contingency tables using the chi-square test of association and Fisher's exact test, when applicable. The risk ratio (RR) will be calculated as a relative risk measure for the primary and secondary outcomes, with a 95% confidence interval being determined. The numbers necessary to treat and obtain a benefit (NNT) and the number needed to treat and obtain a cure (NNH) and their respective 95% confidence intervals will still be calculated.

Regarding the continuous quantitative variables with dissimilar variances, if they present a normal distribution, the comparison between the groups will be performed with Student's t test for non-paired samples (parametric tests). If it is found that the distribution is not normal, the non-parametric Mann-Whitney test will be used. These tests will be used to identify the point differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Low risk patients in active labor admitted to the IMIP; Gestational age between 37 and 42 weeks;
* Cephalic fetus;
* Cervical dilatation up to 8 cm at the time of inclusion in the study.

Exclusion Criteria:

* Indication of cesarean section at the time of the approach;
* Inability to understand and / or perform vocalization maneuvers.
* Patients with Dysphonia
* Deaf and mute patients
* Use of Oxytocin prior to randomization

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
PERINEAL LACERATION Primary outcome: 1. Perineal laceration - present or absent | 1 hour postpartum
  Presence of perineal lacerations observed by the attending staff

SECONDARY OUTCOMES:
DURATION OF SECOND STAGE | 5 hours
  time from complete dilation and delivery
DURATION OF ACTIVE SECOND STAGE | 5 hours
  time from spontaneous pushing to delivery
oxytocin use | 5 hours
  use of oxytocin after randomization
episiotomy | 5 hours
  performance of an episiotomy
instrumental delivery | 5 hours
  use of forceps por vacuum extractor for delivery
laceration degree | 1 hour
  degree of the laceration described by the assistant
Suture need | 4 hours
  need of laceration suturing (including spontaneous lacerations and episiotomies)
Perineal edema | 24 hours
  presence of perineal edema
Maternal satisfaction with the management of the second period | 24 hours
  Maternal satisfaction corresponding to the woman´s impressions and feelings with the management of her second period; evaluated with a scale were women will choose one of the following categories:
  very unsatisfied =1 unsatisfied=2 satisfied=3 very satisfied =4
Perineal pain | 24 hours
  To assess the level of pain a combined scale of pain will be used, and the assessment of this scale meets the visual, categorical, numerical and face scale. The scale varies in discrete numbers from zero to ten, zero being the total absence of pain and ten the most extreme pain that can be felt.
  (67. Chapman CR, Syrjala KL. Measurement of pain. In: Bonica JJ. Pain. 2nd ed. Pennsylvania: Lea & Febiger; 1990:580-94.)
Apgar scores | 5 minutes
  1st and 5th minute Apgar scores recorded in newborns chart
Neonatal ICU admission | 24 hour
  ICU admission need recorded in newborns chart
Need of ressuscitation | 24 hours
  Ressuscitation need recorded in newborns chart

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Neta JN, Amorim MM, Guendler J, Delgado A, Lemos A, Katz L. Vocalization during the second stage of labor to prevent perineal trauma: A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2022 Aug;275:46-53. doi: 10.1016/j.ejogrb.2022.06.007. Epub 2022 Jun 15. PMID 35728488